CLINICAL TRIAL: NCT02170025
Title: Multi-center Phase 2 Study to Assess the Safety, Tolerability and Early Signs of Efficacy of Tid Orally Administered BAY63-2521 in Adult Delta F508 Homozygous Cystic Fibrosis Patients
Brief Title: Early Signs of Efficacy Study With Riociguat in Adult Homozygous Delta F508 Cystic Fibrosis Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated after completion of Part 1, because Part 2 was no longer appropriate.
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17020; 2013-004595-35 (EudraCT Number)
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; delta F508; Safety; Tolerability; Sweat Chloride; Pharmacokinetics
MeSH Terms: conditions — Cystic Fibrosis | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Riociguat (Adempas, BAY63-2521) (Experimental): Participants received 0.5 mg BAY63-2521 three times daily (tid) for 14 days. The dose would be increased to 1 mg BAY63-2521 for an additional 14 days, if this was considered safe and tolerable on the basis of the available data for a given patient.
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)
- Placebo (Experimental): Participants received matching placebo tid.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — Participants received 0.5 mg BAY63-2521 three times daily (tid) for 14 days. The dose would be increased to 1 mg BAY63-2521 for an additional 14 days, if this was considered safe and tolerable on the basis of the available data for a given patient.
  Arms: Riociguat (Adempas, BAY63-2521)
Drug: Placebo — Participants received matching placebo tid.
  Arms: Placebo

SUMMARY:
Assessment of the safety, tolerability and early signs of efficacy of three times a day orally administered BAY63-2521 in adult delta F508 homozygous Cystic Fibrosis patients not on treatment with Orkambi

DETAILED DESCRIPTION:
The study consists of two parts. The first part is double-blind, randomized and placebo-controlled. The second part has an open-label study design. In part 1 patients on Orkambi or other CFTR-modulators are excluded. In part 2 patients on Orkambi are allowed to be included under certain conditions.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent available before any study specific tests or procedures are performed
* Patients must be at least 18 years of age at time of inclusion (i.e. upon signature of informed consent)
* Patient diagnosed with Cystic Fibrosis according to standard criteria (i.e. either elevated sweat chloride content above 60 mmol/ L and/ or genetic testing)
* Patient is homozygous for the deltaF508 mutation
* Patient has a mild-to-moderate stage of lung disease as determined by FEV1 (FEV1 between 40 and 100% predicted)
* Patient has a stable condition of lung disease (no ongoing or recent pulmonary exacerbation and no change in current treatment) within the last 4 weeks prior to screening
* Ability and willingness to understand and follow study procedures for the entire study
* Patients do not smoke. Patients with a history of smoking can be included, if they have refrained from smoking for the last 3 months. If a patients starts smoking during the study participation, he/ she needs to be excluded and considered to be a drop out
* Body mass index (BMI): ≥ 16 kg/ m² (calculated by dividing the patient's weight by the square of his/ her height [kg/ m2])

Inclusion criterion valid for study part 1 only:

- Women of childbearing potential must agree to use adequate contraception when sexually active. 'Adequate contraception' is defined as one highly effective form of contraception (intrauterine devices [IUD], contraceptive implants or tubal sterilization) or a combination of methods (hormone method with a barrier method ). If a partner's vasectomy is the chosen method of contraception or if a partner has documented azoospermia, a hormone or barrier method must be used in combination. Adequate contraception is required from the signing of the informed consent form up until 4 weeks after the last study drug administration

Inclusion criteria valid for study part 2 only:

* Women of childbearing potential must agree to use adequate contraception when sexually active. 'Adequate contraception' is defined as one highly effective form of contraception (intrauterine devices [IUD], contraceptive implants or tubal sterilization) or a combination of methods (hormone method with a barrier method). For patients on Orkambi hormonal methods (including hormonal oral contraceptives) cannot be accepted in this study. They need to choose non-hormonal methods. If a partner's vasectomy is the chosen method of contraception or if a partner has documented azoospermia, a hormone or barrier method must be used in combination. Adequate contraception is required from the signing of the informed consent form up until 4 weeks after the last study drug administration
* Patients receiving Orkambi (Lumcaftor + Ivacaftor) as part of their standard care need to be on stable Orkambi treatment for at least 3 months prior to screening (patients on Lumacaftor and/or Ivacaftor are excluded in part 1)

Exclusion Criteria:

* Patients with Cystic Fibrosis with any background other than homozygous deltaF508 mutation
* Exclusion criterion only valid for study part 1: Patients receiving treatment with Lumacaftor and/ or Ivacaftor
* Active state of hemoptysis or pulmonary hemorrhage, including those events managed by bronchial artery embolization. Also any history of moderate hemoptysis within the 3 months prior to inclusion
* Any history of pneumothorax, bronchial artery embolization or massive hemoptysis. Massive hemoptysis being defined as acute bleeding >240 mL in a 24-hour period or recurrent bleeding >100 mL/ d over several days
* A positive sputum culture for Burkholderia cenocepacia, Burkholderia dolosa, and/ or Mycobacterium abscessus either currently or within the previous year
* Active allergic broncho-pulmonary aspergillosis
* Current pulmonary exacerbation
* Known history of solid organ transplantation
* Known history of any form of pulmonary hypertension
* Clinically relevant deviations of the screened laboratory parameters from reference ranges outside of expected changes for Cystic Fibrosis patients, especially a hemoglobin value below 110 g/L or a creatinine clearance based on the Cockcroft-Gault formula < 15 ml/ min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- United States (3):
  - Birmingham, Alabama
  - Denver, Colorado
  - St Louis, Missouri
- Bruxelles - Brussel, Belgium
- Toronto, Ontario, Canada
- Paris, France
- Berlin, Germany
- Rotterdam, Netherlands
- United Kingdom (2):
  - Belfast, North Ireland
  - London

REFERENCES:
- [Result] Derichs N, Taylor-Cousar JL, Davies JC, Fajac I, Tullis E, Nazareth D, Downey DG, Rosenbluth D, Malfroot A, Saunders C, Jensen R, Solomon GM, Vermeulen F, Kaiser A, Willmann S, Saleh S, Droebner K, Sandner P, Bear CE, Hoffmann A, Ratjen F, Rowe SM; Rio-CF Study Group. Riociguat for the treatment of Phe508del homozygous adults with cystic fibrosis. J Cyst Fibros. 2021 Nov;20(6):1018-1025. doi: 10.1016/j.jcf.2021.07.015. Epub 2021 Aug 19. PMID 34419414
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/17020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multiple centers in 7 countries worldwide between 30-Sep-2014 (first subject first visit) and 31-Jan-2017 (last subject last visit).
Pre-assignment Details: Of 31 participants who were screened, 10 failed screening, 21 were randomized.
Period: Overall Study
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Started | 14 | 7
Completed | 12 | 7
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo | Total
Number analyzed (Participants) | 14 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.1 (6.9) | 29.1 (7.2) | 27.8 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 10 | 6 | 16
Sweat chloride content [Mean (Standard Deviation); unit: mmol/L] — Population: Pharmacodynamic analysis set (N=16) included patients who received the medication and who had valid sweat chloride data for efficacy analysis.
  mmol/L
    number analyzed (Participants) | 9 | 7 | 16
    (all) | 96.33 (17.28) | 94.50 (12.82) | 95.53 (15.03)

OUTCOME MEASURES:

1. Primary Outcome: Change of Sweat Chloride Content From Baseline
Description: Sweat chloride samples were obtained by using a Macroduct induction and collection device according to standard procedures.
Time Frame: Baseline, at day 14 and day 28 in study part 1
Population: Pharmacodynamic analysis set (N=16) included patients who received the medication and who had valid sweat chloride data for efficacy analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 9 | 7
mmol/L
  Change at day 14 in part 1 | 7.06 (10.26) | 8.71 (8.20)
  Change at day 28 in part 1 | 3.44 (11.04) | 9.00 (12.71)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) vs Placebo; Treatment effect describes the difference in outcomes between 0.5 mg riociguat and placebo on Day 14. This was an exploratory analysis. For sample size determination a probabilistic assessment on predicted point estimates and width of credible intervals was performed; Test type: Other; Bayesian analysis = -1.3, 90% CI 2-sided [-8.7 to 6.0]
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) vs Placebo; Treatment effect describes the difference in outcomes between 1.0 mg riociguat and placebo on Day 28. This was an exploratory analysis. For sample size determination a probabilistic assessment on predicted point estimates and width of credible intervals was performed; Test type: Other; Bayesian analysis = -5.0, 90% CI 2-sided [-12.4 to 2.4]

2. Secondary Outcome: Change of FEV1 From Baseline
Description: Spirometry was performed according to the American Thoracic Society Guidelines 1995 at the time points screening/ baseline, treatment period and follow up.
Time Frame: From Baseline to Day 14, Day 28 and Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % predicted value
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 9 | 7
% predicted value
  Change at day 14 | 0.86 (4.59) | 2.00 (7.28)
  Change at day 28 | -0.79 (6.04) | 2.43 (9.55)
  Change at follow-up visit | -0.46 (5.51) | 2.63 (9.50)

ADVERSE EVENTS:
Time Frame: AE events were collected from first treatment until follow up visit 14 days after last treatment
Description: Treatment emergent AEs based on Safety analysis set (N=21)
Arm/Group | Placebo | Riociguat (Adempas, BAY63-2521)
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/14
Other Adverse Events (participants affected / at risk) | 7/7 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | Riociguat (Adempas, BAY63-2521) (N=14)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | Riociguat (Adempas, BAY63-2521) (N=14)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Eye allergy (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Faecal volume decreased (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (3)
Jarisch-Herxheimer reaction (Immune system disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 (2) | 2 (2) — One of these patients had a SAE, which was later downgraded to an AE, and hence is included in both of the tables (Serious AEs and Other AEs).
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1)
Pseudomonas test positive (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (4) | 3 (4)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Based on multiple factors, the design of part 2 is no longer appropriate. Study was terminated at the end of part 1. No safety concerns were identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI(s) shall provide to Bayer any proposed publication or oral presentation relating to the Study or the Study Drug or the Results at least sixty (60) days prior to the intended submission or presentation of the Publication in order to allow Bayer to review it.